# **Informed Consent Form**

Title: Analgesic Effects of Intranasal Diclofenac Sodium, Ibuprofen, and Paracetamol in Pediatric Tonsillectomy Cases

Document Date: 11/12/2024

NCT Number: NCT06731556

Unique Protocol ID: 20.08.2021-E.28962

Purpose of the Study:

This study evaluates the effectiveness and safety of intranasal diclofenac sodium, ibuprofen, and paracetamol for pain management in pediatric tonsillectomy patients.

## Procedures:

- Your child may be placed in one of four groups to receive either intranasal or intravenous pain medication.
- Pain levels will be assessed periodically post-surgery.

### Risks and Benefits:

- Minimal risks are associated with the intranasal drugs.
- Expected benefits include better pain management with fewer side effects.

**Voluntary Participation:** 

- Participation is entirely voluntary, and you may withdraw at any time without affecting your child's treatment.

## Confidentiality:

- All information will be kept confidential.

#### Contact Information:

For any questions, please contact Prof. Dr. Alper Yenigün at alperyenigün@gmail..com or +90 (505) 504 06 96